CLINICAL TRIAL: NCT05672043
Title: Perspective Study on Genetic Predispositions and Clinical Prognosis of Children and Adolescents With Malignant Brain Neoplasms in China
Brief Title: Genetic and Molecular Risk Profiles of Pediatric Malignant Brain Tumors in China
Acronym: GRIPP
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20221226
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Medulloblastoma; Central Nervous System Tumor, Pediatric; Ependymoma; Germ Cell Tumor; Glioma; Brain Tumor, Pediatric
Keywords: medulloblastoma; pediatric brain tumor
MeSH Terms: conditions — Medulloblastoma; Central Nervous System Neoplasms; Ependymoma; Neoplasms, Germ Cell and Embryonal; Glioma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood sample; tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary malignant central nervous system (CNS) tumors are the second most common childhood malignancies. Amongst, medulloblastomas are the most common malignant brain tumor of childhood and occur primarily in the cerebellum. According to molecular characteristics, medulloblastomas were classified into four subtypes: WNT, SHH, Group3 and Group4 and different prognosis were noticed between subgroups. Several genetic predispositions related to clinical outcome were also discovered and might influence the treatment of medulloblastomas as novel pharmaceutical targets. This study aims to investigate genetic and cellular profiles of pediatric brain malignancies, mostly medulloblastomas, and other central nervous system tumor based on WGS, RNA-seq, single-cell sequencing and spatial transcriptomics. We also aim to investigate the correlation between genetic characteristics and clinical prognosis.

DETAILED DESCRIPTION:
This is an observational study including pediatric patients with medulloblastomas, and other central nervous system tumor who are eligible for surgical tumor resection.

Patients will be registered after histological diagnosis is made and meet the inclusion criteria. Epidemiological, histological and radiological information will be collected and Case report form (CRF) will be filled up by investigators. Patients will be follow up 3 months, 6 months, 1 year after surgery and every year afterwards by phone and at clinics. MRI contrast scans are required for each follow-up to assess progression, relapse or metastasis. Patients' neurological status and quality of life will be evaluated during follow-up.

Blood samples and tumor tissue will be collected during surgery. After registry, samples will be send for WGS, whole transcriptome resequencing, single-cell sequencing and spatial transcriptomics as appropriate. Clinical outcome and genetic profiles will be analyzed as appropriate to find out the potential pathogenic factors.

Medulloblastomas samples will be used for culturing primary cells and generating patient-derived xenografts in mice. The latter will be used for in vivo experiments of medulloblastoma pathophysiological mechanisms and pharmaceutical investigations.

ELIGIBILITY:
Inclusion Criteria:

- Children and adolescents aged between 0-18 years old, diagnosed with medulloblastoma or other malignant central nervous system tumors including glioma, ependymoma, germ cell tumors,tuberous sclerosis, neuronal and neuronoglial tumors, choroid plexus tumors, atypical teratoid/rhabdoid tumors, ependymoblastoma, and medulloepithelioma;

Patients must be eligible for and receive tumor resection;

Histological examination by institutional neuro-pathological evaluation must confirmed the diagnosis of brain malignancies;

Participants consent with joining the current study and comply with follow-up visits;

The patients must have no previous radiotherapy or chemotherapy other than corticosteroids.

Exclusion Criteria:

- Patients with major perioperative complications which lead to significant and sudden deterioration;

Patients with major systemic illness (e.g., serious infection or significant cardiac, pulmonary, hepatic, or other organ dysfunction) which might compromise the patient's ability to tolerate standard treatment or would likely interfere with overall prognosis;

Patients with major adverse events or sudden deterioration irrelevant to the current study;

Quality of tumor tissue sample did not meet the criterion for genetic sequencing and laboratory investigations;

Patients who refuse to participate in the study or who request dropping out from the study

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents aged between 0-18 years old, diagnosed with medulloblastoma or other malignant central nervous system tumors in participated institutions in mainland China, with available clinical records and tumor samples, fitting eligibility criteria, are enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years

SECONDARY OUTCOMES:
Progression free survival | 5 years
  No sign of tumor relapse, metastasis or progression confirmed by MRI contrast examination during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hosiptal, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided